CLINICAL TRIAL: NCT05710952
Title: Impact of Orthodontic Treatment on the Temporomandibular Joints (TMJ) Assessed by Modjaw in Adults
Brief Title: Impact of Orthodontic Treatment on the Temporomandibular Joints (TMJ) Assessed by Modjaw
Acronym: EMDJW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL22_0509
Record Dates: First submitted 2023-01-12; First posted 2023-02-02 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Temporomandibular joint; Orthodontic; Modjaw; Orthodontic braces
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Braces (Other): Patients will receive an orthodontic treatment with fixed braces for 12 to 24 months
  Interventions: Device: Review by Modjaw

INTERVENTIONS:
Device: Review by Modjaw — A review by Modjaw's will be done before the braces treatment and after.

SUMMARY:
The aim of the study is to assess the correlation between orthodontic treatment and temporomandibular joint (TMJ). For that, an evaluation with a virtual articulator (Modjaw) is carried out before and after the treatment. The condylar course are compared. Furthermore, the eventual TMJ symptoms are also compared before and after.

ELIGIBILITY:
Inclusion Criteria:

* Major patient (≥18 years)
* First dentofacial orthopedic consultation at the dental clinic of Montpellier
* Patient requiring multi-attachment orthodontic treatment (vestibular or lingual) for a duration ≤2 years
* Signed informed consent

Exclusion Criteria:

* Syndromic patient
* Orthodontic treatment with aligners
* General joint or bone pathology
* Patients with oral hygiene incompatible with orthodontic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2026-04-07 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Gap reduction between the interincisive point in mouth opening and the ordinate axis | Up to 24 months
  Define if there is an improvement in the straightness of the condylar path by measuring the gap between the interincisive point in mouth opening and the ordinate axis in mm assessed by Modjaw

SECONDARY OUTCOMES:
Condylar courses homogeneity | Up to 24 months
  Qualitative comparison of the homogeneity of the condylar courses before and after treatment
Condylar courses symmetry | Up to 24 months
  Qualitative comparison of the symmetry of the condylar symmetry before and after treatment
Condylar courses straightness | Up to 24 months
  Qualitative comparison of the straightness of the condylar symmetry before and after treatment
Amplitude of the condylar path | Up to 24 months
  Virtual path length in mm assessed by Modjaw
Straightness of the condylar path | Up to 24 months
  Y-axis deviation in mm assessed by Modjaw
Adverses events | Up to 24 months
  Adverse events will be assessed before and after treatment
Pain assessment | Up to 24 months
  Pain is assessed by an analogic visual scale from 0 (no pain) to 10 (maximum pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de soins dentaires, Montpellier, France